CLINICAL TRIAL: NCT04871516
Title: A Single Center Phase II Prospective Clinical Trial to Assess the Feasibility of Preoperative Radiation Boost in Breast Cancer Patients
Brief Title: Radiation Therapy Boost Before Surgery for the Treatment of Non-metastatic Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bruce G Haffty, Professor and Chairman, Department of Radiation Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020001306; NCI-2020-05711 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2020001306; 042005 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2021-05-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Invasive Breast Carcinoma; Non-Metastatic Breast Carcinoma; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (radiation therapy boost, WBI) (Experimental): Prior to surgery, patients undergo radiation therapy boost over 4 fractions. Patients then undergo standard of care surgery 1-3 weeks from the last day of boost. 3 to 5 weeks after surgery, patients continue standard of care WBI in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Boost; Procedure: Therapeutic Surgical Procedure; Radiation: Whole Breast Irradiation; Other: Breast MRI

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Boost — Undergo radiation therapy boost
  Other Names: Boost Radiation; Boost Radiation Therapy; Boost Radiotherapy; Radiation Therapy Boost; Radiotherapy Boost
Procedure: Therapeutic Surgical Procedure — Undergo standard surgery
Radiation: Whole Breast Irradiation — Undergo standard WBI
Other: Breast MRI — A baseline breast MRI

SUMMARY:
This phase II trial investigates the safety of delivering a part (boost) of radiation treatment before breast surgery in treating patients with breast cancer that has not spread to other places in the body (non-metastatic). Radiation therapy uses high energy photons/electrons to kill tumor cells and shrink tumors. Delivering a boost radiation treatment before surgery when doctors can still visualize the tumor on imaging may help to better target the tumor and decrease the volume of normal irradiated tissue. By so doing, doctors may achieve better cosmetic outcomes and possibly better tumor control.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that the incidence of grade 3 or more wound complications in patients with non-metastatic node negative breast cancer who are eligible for breast conserving surgery (BCS) and treated with pre-operative radiation boost at 1 month after end of whole breast radiation is no worse than the rates in the current standard of care (6-20%).

SECONDARY OBJECTIVE:

I. To demonstrate that the physician reported cosmetic outcome at 1 and 3 years after the end of treatment is better than what has been reported for the current standard of practice for patients undergoing BCS and hypofractionated whole breast irradiation (WBI).

TERTIARY/EXPLORATORY OBJECTIVES:

I. To measure the acute and late radiation related toxicities such as radiation dermatitis, telangiectasia and fibrosis in this cohort of patients.

II. To measure the pre-operative boost clinical target volume (CTV) and compare to the post-op CTV volume that would have been contoured as CTV if the boost was to be delivered post-operatively.

III. To measure the incidence of fair/poor patient reported cosmetic outcome using the Breast Cancer Treatment Outcomes Scale (BCTOS) cosmetic scale.

IV. To study the cancer biology before and after radiation treatment.

OUTLINE:

Prior to surgery, patients undergo radiation therapy boost over 4 fractions. Patients then undergo standard of care surgery 1-3 weeks from the last day of boost. 3 to 5 weeks after surgery, patients continue standard of care WBI in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, 12, 18, and 24 months

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with biopsy proven invasive cancer
* Clinically and radiographically node negative
* No indication of metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Synchronous bilateral invasive cancer allowed
* Negative serum pregnancy test within one month from the radiation therapy (RT) boost delivery
* Willingness to participate in the clinical trial and adhere to the study protocol
* Individuals of all races, genders and ethnic groups are eligible for this trial

Exclusion Criteria:

* Need for neoadjuvant chemotherapy
* Inflammatory breast cancer (cT4)
* Multicentric tumor
* Prior ipsilateral breast or thoracic RT
* Contraindication for baseline magnetic resonance imaging (MRI)
* Contraindication for surgery
* Distant metastatic disease
* Other synchronous cancer (besides bilateral breast)
* Contraindication to radiation therapy (presence of scleroderma or other collagen vascular disease)
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2027-12-05 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in wound status from baseline every 3-6 months after WBI to access incidence of grade 3 or more wound complications after breast conserving surgery. | For at least 36 months after WBI
  Wound complications will be assessed by the surgeon and radiation oncologist and graded using descriptions and grading scales found in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 5 (CTCAE v 5.0). This will be calculated as a proportion based on the number of events in the study. Will report the proportion with a 95% confidence interval (CI) using the Clopper-Pearson method.

SECONDARY OUTCOMES:
Physician reported cosmesis | At 1 month after whole breast irradiation (WBI)
  Physician reported cosmesis will be assessed using the Harvard Cosmesis assessment Scale for Breast Cancer Patients which is a 4-point scale describing the breast cosmetic outcome (excellent, good, fair or poor).
Physician reported cosmesis | At 12 months after WBI
  Physician reported cosmesis will be assessed using the Harvard Cosmesis assessment Scale for Breast Cancer Patients which is a 4-point scale describing the breast cosmetic outcome (excellent, good, fair or poor).
Physician reported cosmesis | At 36 months after WBI
  Physician reported cosmesis will be assessed using the Harvard Cosmesis assessment Scale for Breast Cancer Patients which is a 4-point scale describing the breast cosmetic outcome (excellent, good, fair or poor). Will be reported as a proportion; CI will be calculated using the Clopper-Pearson model.

OTHER OUTCOMES:
Acute and late radiation toxicity | Up to 24 months after WBI
  Rate of fibrosis, rate of telangiectasia formation and rate of radiation dermatitis will be assessed by the radiation oncologist using descriptions and grading scales found in the NCI CTCAE v5.0. Will also assess changes in pathology between the biopsy and the surgical specimen.
Patient reported cosmesis | At 1 month after WBI
  Patient reported cosmesis will be assessed by the patient using the Breast Cancer Treatment Outcomes Scale (BCTOS).
Patient reported cosmesis | At 12 months after WBI
  Patient reported cosmesis will be assessed by the patient using the Breast Cancer Treatment Outcomes Scale (BCTOS).
  Breast Cancer Treatment Outcome Scale is a questionnaire designed to assess women's subjective evaluation of both the aesthetic and functional outcome after breast cancer treatment. Patients are instructed to rate each item of the BCTOS questionnaire on a four-point scale evaluating the differences between the treated and the untreated breast (1 = no difference to 4 = large difference). Higher scores reflect worse outcomes.
Patient reported cosmesis | At 24 months after WBI
  Patient reported cosmesis will be assessed by the patient using the Breast Cancer Treatment Outcomes Scale (BCTOS).
  Breast Cancer Treatment Outcome Scale is a questionnaire designed to assess women's subjective evaluation of both the aesthetic and functional outcome after breast cancer treatment. Patients are instructed to rate each item of the BCTOS questionnaire on a four-point scale evaluating the differences between the treated and the untreated breast (1 = no difference to 4 = large difference). Higher scores reflect worse outcomes.
Clinical target volume (CTV) | Measured 1-5 weeks prior to surgery and measured 1-7 weeks after surgery
  The difference between the pre-operative boost Clinical target volume (CTV) and the post-op Clinical target volume (CTV) volume that would have been contoured as Clinical target volume (CTV) if the boost was to be delivered post-operatively.
Tumor histology and pathologic response | Up to 24 months after WBI
  Another goal is to look into the histopathology of tumors before and after radiation to assess response and other immunologic changes to the tumor and the tumor environment elicited by the radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G Haffty, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (11):
- United States (11):
  - Clara Maass Medical Center, Belleville, New Jersey
  - RWJBarnabas Health-Trinitas Hospital and Comprehensive Care, Elizabeth, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - RWJBarnabas Health Jersey City Medical Center, Jersey City, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Cooperman Barnabas Medical Center (Saint Barnabas Medical Center), Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT04871516/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT04871516/ICF_001.pdf